CLINICAL TRIAL: NCT07307157
Title: Head-to-Head Evaluation of the Cancer Ontology Supervised Multimodal Orchestration (COSMO) AI System Versus Pathologist-Only Review
Acronym: COSMO
Status: Enrolling by invitation | Type: Observational
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Kun-Hsing Yu, Associate Professor, Harvard Medical School (HMS and HSDM)
Other Study IDs: Yu Lab COSMO Study
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Brain Cancer; Lung Cancer (Diagnosis); Renal Cancer
Keywords: Artificial Intelligence; Whole-Slide Images; Ontology; Multimodal
MeSH Terms: conditions — Brain Neoplasms; Lung Neoplasms; Disease; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AI-Based Evaluation using COSMO
- Pathologist-Based Evaluation
  Interventions: Diagnostic Test: Digital Pathology Evaluation

INTERVENTIONS:
Diagnostic Test: Digital Pathology Evaluation — Digital Pathology Evaluation
  Groups: Pathologist-Based Evaluation

SUMMARY:
This study evaluates the diagnostic performance of the Cancer Ontology Supervised Multimodal Orchestration (COSMO) AI system for cancer subtype classification and compares it head-to-head with pathologist-only review. Pathologists will independently review de-identified whole-slide images derived from up to 300 patients across three anatomical sites (brain, lung, kidney) and provide diagnostic assessments. In parallel, COSMO will process the same cases offline to generate independent predictions, enabling direct comparison of diagnostic accuracy between human experts and the AI system.

The study will characterize the diagnostic accuracy of COSMO and pathologists, inter-observer agreement, and variations in performance across anatomical sites and cancer types with different incidence rates. Results will establish how COSMO compares to pathologists on identical cases and will inform the development of AI-assisted diagnostic systems in clinical practice.

DETAILED DESCRIPTION:
Study Rationale and Background Diagnostic accuracy in cancer subtype classification varies significantly among pathologists due to differences in expertise, experience, and access to diagnostic resources. The emergence of AI systems in pathology offers the potential to enhance diagnostic performance and consistency in cancer classification. However, direct empirical comparisons of AI-based predictions and pathologists' diagnostic performance on identical cases remain limited in the literature.

Study Aims This head-to-head comparative study aims to: (1) evaluate the diagnostic performance of the COSMO AI system in cancer subtype classification across multiple anatomical sites; (2) characterize the diagnostic accuracy of experienced pathologists on the same cases; (3) directly compare diagnostic performance metrics between COSMO and pathologists; and (4) examine concordance patterns and performance variation by anatomical site, cancer incidence category, pathologist experience, and case complexity.

Study Setting and Participants The study will involve up to 25 board-certified pathologists with 3 to 10+ years of diagnostic experience, recruited from institutions across North America, Europe, and the Asia-Pacific region. Participating pathologists will have domain expertise in neuropathology, pulmonary pathology, urologic pathology, or general anatomical pathology.

Cases and Stratification The study will employ de-identified archival whole-slide images representing up to 300 patients with confirmed reference diagnoses, including 100 brain cancers, 100 lung cancers, and 100 kidney cancers. Cases will be stratified by cancer type and incidence category (common vs. rare or uncommon), consistent with World Health Organization (WHO) guidelines.

Data Collection Pathologists will independently review each case and provide diagnostic classifications along with confidence assessments using a 5-point scale. The digital pathology interface will automatically record time-to-diagnosis metrics. COSMO will process the same cases offline to generate independent diagnostic predictions and confidence scores. Both pathologist and AI predictions will be evaluated against established reference standard diagnoses.

Analysis Framework The primary analysis will characterize diagnostic performance metrics (including accuracy, sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and area under the receiver operating characteristic curve (AUROC)) for both pathologists (at the individual and aggregated levels) and the COSMO system. Secondary analyses will assess performance stratified by anatomical site, cancer incidence category, and pathologist experience level.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified pathologist with expertise in neuropathology, pulmonary pathology, urologic pathology, or general anatomical pathology
* Minimum of 3 years of clinical diagnostic experience
* Active clinical practice involving diagnostic pathology slide review
* Willingness to independently review and diagnose up to 300 de-identified whole-slide images
* Ability to access the study platform and complete case reviews within the specified study timeline
* Provision of informed consent for study participation

Exclusion Criteria:

* Prior involvement in the design or validation of the COSMO AI system
* Inability to commit sufficient time to complete assigned case reviews
* Presence of significant financial conflicts of interest related to the study outcomes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will recruit pathologists from international academic medical centers, hospital systems, and diagnostic pathology practices across North America (United States), Europe (Austria, Hungary), and the Asia-Pacific (Taiwan, Hong Kong, South Korea, China, India) region. Participating sites will include major academic institutions with established pathology departments, with recruitment targeting expertise in neuropathology, pulmonary pathology, and urologic pathology.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | Periprocedural (at the time of slide review)
  Diagnostic performance of the COSMO AI system and pathologists in identifying cancer subtypes across brain, lung, and kidney tumors, as assessed by accuracy, balanced accuracy, sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and area under the receiver operating characteristic curve (AUROC). We will include both overall comparisons and stratified evaluations by anatomical site and cancer incidence category (common vs. rare or uncommon).

SECONDARY OUTCOMES:
Inter-Observer Agreement Among Pathologists | Periprocedural (at the time of slide review)
  Diagnostic concordance among participating pathologists, measured by Fleiss' kappa, intraclass correlation coefficient (ICC), and pairwise concordance rates.
Pathologist-COSMO AI Concordance | Periprocedural (at the time of slide review)
  Agreement patterns between pathologist diagnoses and COSMO AI predictions, including proportion of concordant cases overall and stratified by anatomical site, cancer incidence category, and pathologist experience level.
Diagnostic Confidence | Periprocedural (at the time of slide review)
  Mean confidence scores (5-point scale) reported by pathologists during diagnostic assessment, stratified by anatomical site, cancer incidence category, and diagnostic correctness (correct vs. incorrect).
Time-to-Diagnosis | Periprocedural (at the time of slide review)
  Mean diagnostic time (in seconds) required by pathologists to provide cancer subtype classification, stratified by anatomical site, cancer incidence category, and pathologist experience level.
Diagnostic Performance Stratified by Pathologist Experience | Periprocedural (at the time of slide review)
  Diagnostic accuracy of pathologists stratified by years of clinical experience (3-5 years, 6-10 years, >10 years) to assess the relationship between experience level and diagnostic performance in cancer subtype classification.

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Hsing Yu, MD, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Harvard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual pathologist diagnostic assessments will not be shared to protect evaluator anonymity and privacy. De-identified case data and aggregated performance metrics will be made available through published results and supplementary materials. The protocol document will be uploaded to enable full methodological transparency.